CLINICAL TRIAL: NCT01700218
Title: Integrated Telemonitoring and Nurse Support Evaluation in Heart Failure
Brief Title: Integrated Telemonitoring and Nurse Support Evaluation
Acronym: INTENSE-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Collaborators: Ludwig Boltzmann Institute for translational heart failure research (Unknown); AIT Austrian Institute of Technology GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-537 ex 11/12
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Heart Failure
Keywords: telemonitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- telemonitoring (Other): patients in the telemonitoring arm will record vital parameters (blood pressure, heart rate, body weight) and transmit these parameters together with wellbeing and daily dose of heart failure medication
  Interventions: Other: telemonitoring
- control (Other): patients in the control arm will not record any vital parameter
  Interventions: Other: control

INTERVENTIONS:
Other: telemonitoring
  Arms: telemonitoring
Other: control
  Arms: control

SUMMARY:
The purpose of the study is to test a new medical device for optimizing treatment of heart failure and compare its effect on outcome of patients with a recent hospitalization for worsening heart failure

DETAILED DESCRIPTION:
Patients after an episode of acute heart failure have an increased risk of rehospitalisation and impaired prognosis for survival. Neither a sole mobile nurse support nor a sole telemonitoring system has been able to provide consistent data on a beneficial influence on prognosis. Furthermore, the influence of frequent measurements of NT-pro-BNP in a home setting of heart failure patients has not been investigated so far.

This study will test a new medical device (software) for optimizing treatment of heart failure patients and evaluate its impact on outcome of these patients.

ELIGIBILITY:
Inclusion Criteria:

* acute systolic heart failure with admission for at least 4 consecutive days
* treatment with an ACE-inhibitor/angiotensin receptor blocker, beta-blocker, mineralocorticoid receptor antagonist according to current ESC-guidelines
* treatment with a loop diuretic
* stable renal function (eGFR according to MDRD of at least 30ml)
* written informed consent
* minimum age of 18 years

Exclusion Criteria:

* unstable coronary artery disease with revascularisation of any type within the last two months
* planned revascularisation or operation for valvular heart disease within the next 6 months
* planned heart transplantation
* uncontrolled hypertension
* active myocarditis
* malignant disease with a life expectancy of less than 18 months
* chronic use of high-dose NSAID or COX-2-inhibitors
* psychiatric disorders that make it unlikely to understand the protocol
* participation in an other randomized trial
* inability to operate a smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-04 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
all cause mortality and hospitalization for worsening heart failure | 12 months
  outcome assessment will be done by a blinded committee

SECONDARY OUTCOMES:
days alive and out of hospital | 12 months

OTHER OUTCOMES:
exploratory endpoint | 12 months
  The exploratory endpoint will focus on the percentage of optimal dosing (according to current ESC-guidelines) for ACE-inhibitors, angiotensin receptor blockers and beta-blockers

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich M Fruhwald, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University, Graz, Austria